CLINICAL TRIAL: NCT02033980
Title: Efficacy of NICE Classification in the Histological Evaluation of Colorectal Lesions ----- a Multicenter Study in China
Brief Title: Efficacy of NICE Classification in the Histological Evaluation of Colorectal Lesions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: Changhai Hospital (Other); Peking University People's Hospital (Other); Peking Union Medical College Hospital (Other); Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Zhizheng Ge, Ren Ji Hospital, School of medicine, Shanghai Jiao Tong University, Shanghai Jiao Tong University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: rjxh[2013]125
Record Dates: First submitted 2013-12-27; First posted 2014-01-13 (Estimated); Last update posted 2016-05-10 (Estimated); Status verified 2016-05

CONDITIONS: Colorectal Polyps
Keywords: narrow band imaging(NBI); NICE classification; colorectal lesions; predicting histology

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- colorectal lesions (Other): All lesions will be observed with NBI and removed endoscopically or surgically for histological diagnosis.
  Interventions: Device: NBI

INTERVENTIONS:
Device: NBI — All detected colorectal lesions will be examined by high-definition NBI. For type 2 and type 3 lesions, subsequent magnifying NBI examination will be performed.
  Other Names: Evis Lucera system (CV-260, Olympus Inc, Japan); high-definition colonoscopes (CF-H260AL, Olympus Inc, Japan); magnifying colonoscopes (CF-H260AZL, Olympus Inc, Japan)

SUMMARY:
Recently, a new category classification (NICE classification) using non-magnified NBI has been proposed. We design this multicenter study to evaluate the reliability and validity of the NICE classification in diagnosing colorectal polyps by Chinese endoscopists during both image and real-time process.

DETAILED DESCRIPTION:
Many reports have demonstrated the efficacy of narrow band imaging (NBI) with magnification in predicting the histology and invasion depth of colorectal polyps. In China, however, the magnifying endoscope is not used in some medical centers. Even in centers equipped with this technique, the magnifying colonoscope is not sufficiently used in daily practice. Recently, a simple category classification (NICE classification) using non-magnified NBI has been proposed, which classifies colorectal tumors into types 1-3 based on different characteristics of color, surface pattern, and microvessels. Type-1 is considered an index for hyperplastic lesions, type-2 is an index for adenoma or mucosal/SM scanty invasive carcinoma and type-3 is an index for deep SM invasive carcinoma. The new classification has soon arouse attention and been validated in some centers on the efficacy of differentiating adenomatous and hyperplastic polyps. However, most studies enrolled diminutive polyps less than 5mm and the efficacy of non-magnified NBI in differentiating type-2 and type-3 lesions has not been reported. To promote this simple classification, we design this multicenter study to evaluate the predictive validity and performance characteristics of the non-magnified NBI in diagnosing polyps during both image and real-time process.

ELIGIBILITY:
Inclusion Criteria:

* Patients with colorectal lesions during colonoscopy examination
* Informed consent available

Exclusion Criteria:

* Suspect of advanced colorectal cancer
* History of colorectal surgery, familial adenomatous polyposis or inflammatory bowel disease
* Poor bowel preparation
* Patients under unsuitable conditions for examination or treatment, such as acute upper gastrointestinal bleeding, noncorrectable coagulopathy, severe systemic disease, etc

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2016-05; Primary Completion 2017-06 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Accuracy of NICE classification in histological prediction by gastroenterological fellows | within two weeks after polypectomy
  Diagnostic accuracy of gastroenterological fellows using non-magnified NBI according to NICE classification in histological prediction of polyps, compared with histologic examination

SECONDARY OUTCOMES:
Diagnostic accuracy of high-definition and magnifying NBI for type 2 and type 3 lesions. | two weeks after endoscopical or surgical resection
  For lesions identified as type 2 or type 3, subsequent magnifying NBI examination will be performed by NBI experts. Before that, experts will make their own assessment according to all the images taken by gastroenterological fellows, blind to their diagnosis. Then experts will examine the lesions using magnifying endoscopy with NBI capability and make a new assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Zhizheng Ge, MD,Ph.D, Principal Investigator — Renji Hospital, School of Medicine, Shanghai Jiaotong University, Shanghai ,China.
Locations (1):
- Ren Ji Hospital, School of Medicine, Shanghai Jiaotong University, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zhang QW, Zhang JJ, Yang AM, Sheng JQ, Liu YL, Li ZS, Chen HY, Feng N, Jiang QW, Jin P, Zhang LM, Fu HY, Gao YJ, Ge ZZ, Li XB. Feasibility of using narrow band imaging international colorectal endoscopic classification for diagnosing colorectal neoplasia in China: A multicenter pilot observational study. J Dig Dis. 2020 Feb;21(2):88-97. doi: 10.1111/1751-2980.12841. PMID 31895484